CLINICAL TRIAL: NCT00478933
Title: Diagnostic Data Influence on Disease Management and Relation of Genetic Polymorphisms to Tachy-arrhythmia in ICD Patients.
Brief Title: DISCOVERY: Diagnostic Data and Genetic Polymorphisms in ICD Patients.
Acronym: DISCOVERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: DISCOVERY
Record Dates: First submitted 2007-05-23; First posted 2007-05-25 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2017-07

CONDITIONS: Death, Sudden, Cardiac; Ventricular Fibrillation; Tachycardia; Atrial Fibrillation; Sick Sinus Syndrome
Keywords: Arrhythmia; Ventricular; Atrial; Tachycardia; Fibrillation; Flutter; GNB3; GNAS; GNAQ
MeSH Terms: conditions — Death, Sudden, Cardiac; Ventricular Fibrillation; Tachycardia; Atrial Fibrillation; Sick Sinus Syndrome; Arrhythmias, Cardiac | interventions — Defibrillators; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: patients and investigators were blinded to the genetic markers during the study. Therefore, no arm is specified as this is not applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICD Therapy, blood sampling (Experimental): Blood sampling Defibrillator, Dual Chamber ; Implantable
  Interventions: Device: Defibrillator, Dual Chamber ; Implantable; Procedure: Blood sampling

INTERVENTIONS:
Device: Defibrillator, Dual Chamber ; Implantable — Patient must wear a dual chamber ICD to remain in study. Can be enrolled 10 days prior to implant. Is excluded if device type changes.
Procedure: Blood sampling — Blood sampling

SUMMARY:
To prospectively evaluate if the analysis of genetic polymorphisms can be used to identify patients at risk of ventricular tachycardia.

To evaluate the influence of ICD-based diagnostic information on the long term treatment and management of primary prevention ICD-patients.

DETAILED DESCRIPTION:
Evaluate the positive predictive value of single nucleotide polymorphisms (SNPs) in the genes GNB3, GNAS and GNAQ as predictors of ventricular arrhythmia <400 msec.

1. Evaluate the positive predictive value of Single Nucleotide Polymorphisms as predictor for death, cardiac death and atrial fibrillation/flutter in the genes GNB3, GNAS, GNAQ and other SNPs involving signal transduction components which impact on the activity of cardiac ion channels.
2. Evaluate the best combination of genetic parameters, baseline data and follow-up data as predictor of primary endpoint, All cause Mortality, cardiac death and atrial arrhythmia.
3. Evaluate the usage of ICD-system diagnostics (battery status, impedance, pacing threshold, sensing) resulting in medical consequences*.
4. Evaluate the usage of ICD-based patient diagnostics (arrhythmia, IEGM, heart frequency, %pacing, Cardiac Compass) resulting in medical consequences*.
5. Evaluate the frequency of programming changes involving AF-prevention and AF-therapy algorithms.
6. Evaluate the frequency of pacing-parameter programming changes and the resulting medical consequences*.

   * Medical consequences include: Hospitalization, medical interventions, medication, surgery, additional diagnostics and ICD-programming changes.

ELIGIBILITY:
Inclusion Criteria:

* Implantation of a market approved Medtronic Dual-chamber ICD with long term clinical trends Cardiac Compass,
* Subjects requiring the implantation of an ICD for primary prevention according to the current AHA/ACC/ESC guidelines,
* Subject able to comply with the Clinical InvestigationPlan,
* Subject is expected to remain available for follow-up visits,
* Subject has signed the informed consent form within 10 days of implant,
* The system implanted for this study is the first ICD implant for patient.

Exclusion Criteria:

* Women who are pregnant, or women of childbearing potential not on a reliable form of birth control,
* Subject is enrolled in a concurrent study that may confound the results of this study,
* Subject has a life expectancy less than two years,
* Subject is post heart transplant or awaiting heart transplantation,
* Subject is anticipated to demonstrate poor compliance,
* Subjects with syndromes known to be associated with ion channel pathologies such as:

  * Long- or short-QT Syndrome
  * Brugada Syndrome
  * Catecholaminergic Polymorphic Ventricular Tachycardia (CPTV ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1223 (Actual)
Dates: Start 2007-02; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Corrado, MD, Principal Investigator — University of Padova, Italy; Heiner Wieneke, MD, Principal Investigator — Universitätsklinikum Essen, Germany

IPD SHARING:
Plan to Share IPD: No
study is closed several years ago; this is not applicable for this study

REFERENCES:
- [Derived] Wieneke H, Svendsen JH, Lande J, Spencker S, Martinez JG, Strohmer B, Toivonen L, Le Marec H, Garcia-Fernandez FJ, Corrado D, Huertas-Vazquez A, Uy-Evanado A, Rusinaru C, Reinier K, Foldesi C, Hulak W, Chugh SS, Siffert W. Polymorphisms in the GNAS Gene as Predictors of Ventricular Tachyarrhythmias and Sudden Cardiac Death: Results From the DISCOVERY Trial and Oregon Sudden Unexpected Death Study. J Am Heart Assoc. 2016 Nov 28;5(12):e003905. doi: 10.1161/JAHA.116.003905. PMID 27895044

RESULTS

PARTICIPANT FLOW:
Groups:
- ICD Therapy, Blood Sampling: Defibrillator, Dual Chamber ; Implantable: Patient must wear a dual chamber ICD to remain in study. Can be enrolled 10 days prior to implant. Is excluded if device type changes.
  Blood sampling: Blood sampling for genetic analysis of the pre-identified SNPs
Period: Overall Study
Arm/Group | ICD Therapy, Blood Sampling
Started | 1223
Completed | 1145
Not Completed | 78
Not completed — Protocol Violation | 22
Not completed — Informed consent not verified | 3
Not completed — Inadequate data available | 53

BASELINE CHARACTERISTICS:
Groups:
- ICD Therapy, Blood Sampling: Defibrillator, Dual Chamber ; Implantable: Patient must wear a dual chamber ICD to remain in study. Can be enrolled 10 days prior to implant. Is excluded if device type changes.
  Blood sampling: Blood sampling for genetic analysis on pre-specified SNPs
Arm/Group | ICD Therapy, Blood Sampling
Number analyzed (Participants) | 1198
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194
  Male | 1004
Region of Enrollment [Number; unit: participants] — Measures are completed for total enrolled population, including those with inadequate data for analysis.
  participants
    Austria | 40
    Denmark | 57
    Spain | 189
    Finland | 25
    France | 84
    Germany | 491
    Greece | 26
    Hungary | 59
    Italy | 54
    Norway | 26
    Poland | 134
    United Kingdom | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Ventricular Arrhythmia <400 Msec. by GNAS c.393C>T Genotype
Description: The GNAS c.393C>T single nucleotide polymorphism (SNP) was one of seven SNP's analyzed. Patients with de novo ICD implants were genotyped and followed for up to 2 years. All episodes of arrhythmia <400 msec. detected by the device were adjudicated by an independent committee. The number of patients with true arrhythmias <400 msec were tracked by genotype.
Time Frame: 2 years
Measure: Number; unit: participants with VT < 400 msec
Groups:
- c.393C>T CC Genotype: Patients in this group have two copies of the major (C) allele for the c.393C>T single nucleotide polymorphism (SNP) in the GNAS gene
- c.393C>T CT Genotype: Patients in this group have one copy of each allele (C and T) for the c.393C>T single nucleotide polymorphism (SNP) in the GNAS gene
- c.393C>T TT Genotype: Patients in this group have two copies of the minor (T) allele for the c.393C>T single nucleotide polymorphism (SNP) in the GNAS gene
Arm/Group | c.393C>T CC Genotype | c.393C>T CT Genotype | c.393C>T TT Genotype
Number analyzed (Participants) | 285 | 555 | 305
participants with VT < 400 msec | 63 | 136 | 98

2. Secondary Outcome: Hospitalization, Medical Interventions, Medication, Surgery, Additional Diagnostics
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: All Cause Mortality, Cardiac Death and Atrial Fibrillation/Flutter
Time Frame: 2 years
Reporting Status: Not Posted

4. Primary Outcome: Number of Patients With Ventricular Arrhythmia <400 Msec. by GNAS c.2273C>T Genotype
Description: The GNAS c.2273C>T single nucleotide polymorphism (SNP) was one of seven SNP's analyzed. Patients with de novo ICD implants were genotyped and followed for up to 2 years. All episodes of arrhythmia <400 msec. detected by the device were adjudicated by an independent committee. The number of patients with true arrhythmias <400 msec were tracked by genotype.
Time Frame: 2 years
Measure: Number; unit: participants with VT < 400 msec
Groups:
- c.2273C>T CC Genotype: Patients in this group have two copies of the major (C) allele for the c.2273C>T single nucleotide polymorphism (SNP) in the GNAS gene
- c.2273C>T CT Genotype: Patients in this group have one copy of each (C and T) allele for the c.2273C>T single nucleotide polymorphism (SNP) in the GNAS gene
- c.393C>T TT Genotype: Patients in this group have two copies of the minor (T) allele for the c.2273C>T single nucleotide polymorphism (SNP) in the GNAS gene
Arm/Group | c.2273C>T CC Genotype | c.2273C>T CT Genotype | c.393C>T TT Genotype
Number analyzed (Participants) | 456 | 533 | 156
participants with VT < 400 msec | 103 | 136 | 59

5. Primary Outcome: Number of Patients With Ventricular Arrhythmia <400 Msec. by GNAS c.2291C>T Genotype
Description: The GNAS c.2291C>T single nucleotide polymorphism (SNP) was one of seven SNP's analyzed. Patients with de novo ICD implants were genotyped and followed for up to 2 years. All episodes of arrhythmia <400 msec. detected by the device were adjudicated by an independent committee. The number of patients with true arrhythmias <400 msec were tracked by genotype.
Time Frame: 2 years
Measure: Number; unit: participants with VT < 400 msec
Groups:
- c.2291C>T CC Genotype: Patients in this group have two copies of the major (C) allele for the c.2291C>T single nucleotide polymorphism (SNP) in the GNAS gene
- c.2291C>T CT Genotype: Patients in this group have one copy of each allele (C and T) for the c.2291C>T single nucleotide polymorphism (SNP) in the GNAS gene
- c.2291C>T TT Genotype: Patients in this group have two copies of the minor (T) allele for the c.2291C>T single nucleotide polymorphism (SNP) in the GNAS gene
Arm/Group | c.2291C>T CC Genotype | c.2291C>T CT Genotype | c.2291C>T TT Genotype
Number analyzed (Participants) | 527 | 508 | 110
participants with VT < 400 msec | 145 | 123 | 29

6. Primary Outcome: Number of Patients With Ventricular Arrhythmia <400 Msec. by GNAQ c.-909/-908GC>TT Genotype
Description: The GNAQ c.-909/-908GC>TT single nucleotide polymorphism (SNP) was one of seven SNP's analyzed. Patients with de novo ICD implants were genotyped and followed for up to 2 years. All episodes of arrhythmia <400 msec. detected by the device were adjudicated by an independent committee. The number of patients with true arrhythmias <400 msec were tracked by genotype.
Time Frame: 2 years
Measure: Number; unit: participants with VT < 400 msec
Groups:
- GNAQ c.-909/-908GC>TT GC/GC Genotype: Patients in this group have two copies of the major (GC) allele for the c.-909/-908GC>TT single nucleotide polymorphism (SNP) in the GNAQ gene
- GNAQ c.-909/-908GC>TT GC/TT Genotype: Patients in this group have one copy of each allele (GC and TT) for the c.-909/-908GC>TT single nucleotide polymorphism (SNP) in the GNAS gene
- GNAQ c.-909/-908GC>TT TT/TT Genotype: Patients in this group have two copies of the minor (TT) allele for the c.-909/-908GC>TT single nucleotide polymorphism (SNP) in the GNAQ gene
Arm/Group | GNAQ c.-909/-908GC>TT GC/GC Genotype | GNAQ c.-909/-908GC>TT GC/TT Genotype | GNAQ c.-909/-908GC>TT TT/TT Genotype
Number analyzed (Participants) | 342 | 546 | 257
participants with VT < 400 msec | 85 | 143 | 69

7. Primary Outcome: Number of Patients With Ventricular Arrhythmia <400 Msec. by GNAQ c.-382G>A Genotype
Description: The GNAQ c.-382G>A single nucleotide polymorphism (SNP) was one of seven SNP's analyzed. Patients with de novo ICD implants were genotyped and followed for up to 2 years. All episodes of arrhythmia <400 msec. detected by the device were adjudicated by an independent committee. The number of patients with true arrhythmias <400 msec were tracked by genotype.
Time Frame: 2 years
Measure: Number; unit: participants with VT < 400 msec
Groups:
- c.-382G>A GG Genotype: Patients in this group have two copies of the major (G) allele for the c.-382G>A single nucleotide polymorphism (SNP) in the GNAQ gene
- c.-382G>A GA Genotype: Patients in this group have one copy of each allele (C and T) for the c.-382G>A single nucleotide polymorphism (SNP) in the GNAQ gene
- c.-382G>A AA Genotype: Patients in this group have two copies of the minor (A) allele for the c.-382G>A single nucleotide polymorphism (SNP) in the GNAQ gene
Arm/Group | c.-382G>A GG Genotype | c.-382G>A GA Genotype | c.-382G>A AA Genotype
Number analyzed (Participants) | 945 | 189 | 11
participants with VT < 400 msec | 253 | 42 | 2

8. Primary Outcome: Number of Patients With Ventricular Arrhythmia <400 Msec. by GNAQ c.-387G>A Genotype
Description: The GNAQ c.-387G>A single nucleotide polymorphism (SNP) was one of seven SNP's analyzed. Patients with de novo ICD implants were genotyped and followed for up to 2 years. All episodes of arrhythmia <400 msec. detected by the device were adjudicated by an independent committee. The number of patients with true arrhythmias <400 msec were tracked by genotype.
Time Frame: 2 years
Measure: Number; unit: participants with VT < 400 msec
Groups:
- c.-387G>A GG Genotype: Patients in this group have two copies of the major (G) allele for the c.-387G>A single nucleotide polymorphism (SNP) in the GNAQ gene
- c.-387G>A GA Genotype: Patients in this group have one copy of each allele (C and T) for the c.-387G>A single nucleotide polymorphism (SNP) in the GNAQ gene
- c.-387G>A AA Genotype: Patients in this group have two copies of the minor (A) allele for the c.-387G>A single nucleotide polymorphism (SNP) in the GNAQ gene
Arm/Group | c.-387G>A GG Genotype | c.-387G>A GA Genotype | c.-387G>A AA Genotype
Number analyzed (Participants) | 1041 | 101 | 3
participants with VT < 400 msec | 268 | 29 | 0

9. Primary Outcome: Outcome Measure Title: Number of Patients With Ventricular Arrhythmia <400 Msec. by GNB3 c.825C>T Genotype
Description: The GNB3 c.825C>T single nucleotide polymorphism (SNP) was one of seven SNP's analyzed. Patients with de novo ICD implants were genotyped and followed for up to 2 years. All episodes of arrhythmia <400 msec. detected by the device were adjudicated by an independent committee. The number of patients with true arrhythmias <400 msec were tracked by genotype.
Time Frame: 2 years
Measure: Number; unit: participants with VT < 400 msec
Groups:
- c.825C>T CC Genotype: Patients in this group have two copies of the major (G) allele for the c.825C>T CC single nucleotide polymorphism (SNP) in the GNB3 gene
- c.825C>T CT Genotype: Patients in this group have one copy of each allele (C and T) for the c.825C>T single nucleotide polymorphism (SNP) in the GNB3 gene
- c.825C>T TT Genotype: Patients in this group have two copies of the minor (A) allele for the c.825C>T single nucleotide polymorphism (SNP) in the GNB3 gene
Arm/Group | c.825C>T CC Genotype | c.825C>T CT Genotype | c.825C>T TT Genotype
Number analyzed (Participants) | 536 | 499 | 110
participants with VT < 400 msec | 135 | 136 | 26

ADVERSE EVENTS:
Time Frame: From 1st enrollment, 25 April 2007, through last follow up, 31 July 2012: ~ 5 yrs
Description: Only Serious Adverse Device Effects and Serious Procedure-related Adverse Events (in France only) had to be reported.
  Serious Procedure-related Adverse Events (France only): An SAE that occurs due to any procedure specific to the clinical investigation, including the implantation or modification of the system.
Groups:
- ICD Therapy, Blood Sampling: Defibrillator, Dual Chamber ; Implantable: Patient must wear a dual chamber ICD to remain in study. Can be enrolled 10 days prior to implant. Is excluded if device type changes.
  Blood sampling: Blood sampling for genetic analysis on pre-identified SNPs
Arm/Group | ICD Therapy, Blood Sampling
Serious Adverse Events (participants affected / at risk) | 265/1145
Other Adverse Events (participants affected / at risk) | 45/1145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICD Therapy, Blood Sampling (N=1145)
Implant site pain (General disorders) | 1 (1)
Abdominal operation (Surgical and medical procedures) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (3)
aneamia (Blood and lymphatic system disorders) | 1 (1)
angina pectoris (Cardiac disorders) | 5 (8)
aortic aneurysm (Vascular disorders) | 1 (1)
arrhythmia (Cardiac disorders) | 1 (1)
arrhythmia supraventricular (Cardiac disorders) | 1 (1)
arteriogram coronary (Investigations) | 1 (1)
asthenia (General disorders) | 1 (1)
atrial fibrillation (Cardiac disorders) | 11 (13)
atrial flutter (Cardiac disorders) | 1 (1)
atrial tachycardia (Cardiac disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
bile duct stone (Hepatobiliary disorders) | 1 (1)
bradyarrhythmia (Cardiac disorders) | 1 (1)
cardiac ablation (Surgical and medical procedures) | 1 (1)
cardiac failure (Cardiac disorders) | 27 (31)
cardiac failure acute (Cardiac disorders) | 1 (1)
cardiac failure chronic (Cardiac disorders) | 3 (3)
cardiac tamponade (Cardiac disorders) | 1 (1)
cardiogenic shock (Cardiac disorders) | 1 (1)
cardioversion (Surgical and medical procedures) | 1 (1)
cerebellar stroke (Nervous system disorders) | 1 (1)
cerebral infarction (Nervous system disorders) | 1 (1)
cerebrovascular accident (Nervous system disorders) | 3 (3)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
chest discomfort (General disorders) | 1 (1)
chest pain (General disorders) | 4 (4)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
circulatory collapse (Vascular disorders) | 1 (1)
colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Complication associated with device (General disorders) | 1 (1)
cororary artery disease (Cardiac disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
death (General disorders) | 3 (3)
deep venous thrombosis (Vascular disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1)
device dislocation (Product Issues) | 2 (3)
Device electrical impedance issue (Product Issues) | 9 (9)
device extrusion (Product Issues) | 1 (1)
device issue (Product Issues) | 1 (1)
device lead damage (Product Issues) | 2 (2)
device lead issue (Product Issues) | 3 (3)
device malfunction (Product Issues) | 5 (5)
device pacing issue (Product Issues) | 3 (4)
device related infection (Infections and infestations) | 1 (1)
device stimulation issue (Product Issues) | 2 (2)
dizziness (Nervous system disorders) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
gastrointestinal uler haemorrhage (Gastrointestinal disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
gout (Metabolism and nutrition disorders) | 1 (1)
haematoma (Vascular disorders) | 1 (1)
haemorrhage (Vascular disorders) | 1 (1)
heart failure (Cardiac disorders) | 3 (3)
hospitalisation (Surgical and medical procedures) | 3 (4)
hypertension (Cardiac disorders) | 1 (1)
hypertensive nephropathy (Renal and urinary disorders) | 1 (1)
hyperthyroidism (Endocrine disorders) | 1 (1)
hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
ill-defined disorder (General disorders) | 2 (2)
implant site haematoma (General disorders) | 5 (5)
implant site infection (Injury, poisoning and procedural complications) | 7 (7)
implant site infection (Infections and infestations) | 1 (1)
implant site swelling (General disorders) | 1 (1)
implant site ulcer (General disorders) | 1 (1)
inflammatory marker increased (Investigations) | 1 (1)
invertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
ischaemic cardiomayopathy (Cardiac disorders) | 1 (1)
ischaemic stroke (Nervous system disorders) | 1 (1)
lead dislodgement (Product Issues) | 20 (21)
lung infection (Infections and infestations) | 1 (1)
medical device site abscess (Infections and infestations) | 1 (1)
Medical device site extravasation (General disorders) | 1 (1)
multiple injuries (Injury, poisoning and procedural complications) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1)
opthalmic herpes simplex (Infections and infestations) | 1 (1)
orthopnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ovarian cyst (Reproductive system and breast disorders) | 1 (1)
oversensing (Product Issues) | 5 (5)
Pacemaker generated arrhythmia (General disorders) | 1 (1)
pain (General disorders) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
palpitations (Cardiac disorders) | 3 (3)
paroxysmal arrhythmia (Cardiac disorders) | 1 (1)
Peripheral artery stent insertion (Surgical and medical procedures) | 1 (1)
peripheral artery thrombosis (Vascular disorders) | 1 (1)
pneumonia (Infections and infestations) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 (7)
pocket erosion (Injury, poisoning and procedural complications) | 2 (2)
presyncope (Nervous system disorders) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
renal failure (Renal and urinary disorders) | 3 (4)
silent myocardial infarction (Cardiac disorders) | 1 (1)
small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
stent placement (Surgical and medical procedures) | 1 (1)
supraventricular extrasystoles (Cardiac disorders) | 1 (1)
therapy non-responder (General disorders) | 1 (1)
thrombosis (Vascular disorders) | 1 (1)
transient global amnesia (Nervous system disorders) | 1 (1)
traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (2)
undersensing (Product Issues) | 7 (7)
urinary tract infection bacterial (Infections and infestations) | 1 (1)
vena cava thrombosis (Vascular disorders) | 1 (1)
ventricular arrhythmia (Cardiac disorders) | 4 (4)
ventricular fibrillation (Cardiac disorders) | 6 (6)
ventricular tachycardia (Cardiac disorders) | 8 (9)
wound necrosis (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICD Therapy, Blood Sampling (N=1145)
abscess (Infections and infestations) | 1 (1)
acute coronary syndrome (Cardiac disorders) | 1 (1)
acute haemorrhagic ulcerative colitis (Gastrointestinal disorders) | 1 (1)
alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1)
atrial fibrillation (Cardiac disorders) | 3 (3)
cardiac death (General disorders) | 1 (1)
cardiac failure (Cardiac disorders) | 2 (2)
cardiac failure acute (Cardiac disorders) | 1 (1)
cardiac tamponade (Cardiac disorders) | 1 (1)
carpal tunnel syndrome (Nervous system disorders) | 1 (1)
cerebrovascular accident (Nervous system disorders) | 1 (1)
chest pain (General disorders) | 1 (1)
depression (Psychiatric disorders) | 1 (1)
device extrusion (Product Issues) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
dizziness (Nervous system disorders) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1)
hospitalisation (Surgical and medical procedures) | 1 (1)
hypertensive emergency (Vascular disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
implant site haematoma (General disorders) | 1 (2)
implant site infection (Injury, poisoning and procedural complications) | 1 (1)
implant site infection (Infections and infestations) | 1 (1)
implant site pain (General disorders) | 2 (2)
malaise (General disorders) | 1 (1)
Medical device site haematoma (General disorders) | 1 (1)
pneumonia (Infections and infestations) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
presyncope (Nervous system disorders) | 1 (1)
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
sciatica (Nervous system disorders) | 1 (1)
sepsis (Infections and infestations) | 1 (1)
sinus tachycardia (Cardiac disorders) | 1 (1)
sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
spinal pain (Musculoskeletal and connective tissue disorders) | 1 (2)
supraventricular tachycardia (Cardiac disorders) | 1 (1)
ventricular tachycardia (Cardiac disorders) | 2 (2)
wound secretion (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
The following limitations can be noted:

• Patient follow-up was prematurely terminated after at least 12-month follow-up data on all enrolled patients but before the planned 24-month follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days